CLINICAL TRIAL: NCT01221662
Title: Complementary Therapy of Siwu Tang on Patients With Brain Hypoperfusion Syndrome
Brief Title: Efficiency Study of Siwu Tang to Treat Brain Hypoperfusion Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chun-Chung Chen, China Medical University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMR98-IRB-282
Record Dates: First submitted 2010-10-10; First posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Brain Hypoperfusion Syndrome; Ischemia Brain
Keywords: Siwu tang; brain hypoperfusion; cognition function
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Siwu Tang — Siwu Tang 3 g bid(oral) continuously two weeks

SUMMARY:
Brain hypoperfusion patients may cause vascular dementia results from their hypoperfusion state except that is a risk factor for stroke. The most common clinical symptom of hypoperfusion syndrome is dizziness.Siwu tang is made of Angelica sinensis (Oliv.) Diels (當歸), Rehmannia glutinosa (Gaertn) Libosch (熟地黃), Paeonia lactiflora Pall (白芍), Ligusticum chuanxiong Hort (川芎), and that was used to treat patients with blood deficiency for several centuries. the purpose of the present study was to investigate the complementary effect of siwu tang on brain hypoperfusion syndrome patients

DETAILED DESCRIPTION:
We designed a randomized, double-blinded controlled study, and a total of 80 patients with brain hypoperfusion syndrome should be finished assessment in two years. The 80 patients with hypoperfusion syndrome were divided into as follows:1) control group, receiving siwu tang placebo 3 g bid continuously two weeks except ordinary treatment; 2) treatment group, receiving siwu tang 3 g bid continuously two weeks except ordinary treatment. The patients were assessed before, and 4 weeks (weeks±3 days) and 12 weeks (12 weeks±3 days) after siwu tang treatment, respectively. Primary outcome measure was cerebral blood flow by using single photon emission computed tomography (SPECT); Second outcome measure included severity of dizziness by using visual analogue scale (VAS); cognitive function by using Mini-Mental Status (MMSE), Cognitive Abilities Screening Instrument (CASI), and Clinical Dementia Rating (CDR); quality of life by using barthel index (BI) and Functional Independent Measure (FIM).

We predict that siwu tang can improve cerebral blood flow, and clinical manifestation including dizziness, and cognition function and quality of life in patients with brain hypoperfusion syndrome .

ELIGIBILITY:
Inclusion Criteria:

* age between 18y/o to 80 y/o and had brain hypoperfusion syndrome such as dizziness
* barthel index (BI) > 60。
* single photon emission computer tomography(SPECT) or MRI exam show hypoperfusion area

Exclusion Criteria:

* Patient had cancer or uremia,liver cirrhosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
cerebral blood flow | 12 weeks after treatment
  Primary outcome measure was cerebral blood flow by using single photon emission computed tomography (SPECT)

SECONDARY OUTCOMES:
severity of dizziness | 12 weeks after treatment
  severity of dizziness by using visual analogue scale (VAS)
cognitive function | 12 weeks after treatment
  cognitive function by using Mini-Mental Status (MMSE), Cognitive Abilities Screening Instrument (CASI), and Clinical Dementia Rating (CDR)
quality of life | 12 weeks after treatment
  quality of life by using barthel index (BI) and Functional Independent Measure (FIM)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Chung Chen, master, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan